CLINICAL TRIAL: NCT00468897
Title: An Open-Label, Randomized, Two-Period Crossover Study to Demonstrate the Bioequivalence of a Tablet Formulation of Rosiglitazone XR (BRL-049653) 8mg Manufactured at Two Different Sites in Healthy Volunteers in Fasting Conditions
Brief Title: A Study To Demonstrate The Bioequivalence Of Rosiglitazone XR (BRL-049653) 8mgs XR Manufactured At Two Different Sites.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AXR107453
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimers Disease; healthy volunteers; bioequivalence
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm AB (Experimental): A will be a single tablet RSG XR 8 milligram (mg) manufactured in Harlow administered in the fasted state and B will be a single tablet RSG XR 8 mg manufactured in Crawley administered in the fasted state. In Arm AB subject will receive A regimen in Period 1 and B regimen in Period 2.There will be wash-out period of 5 days between doses.
  Interventions: Drug: RSG XR
- Treatment Arm BA (Experimental): A will be a single tablet RSG XR 8 mg manufactured in Harlow administered in the fasted state and B will be a single tablet RSG XR 8 mg manufactured in Crawley administered in the fasted state. In Arm BA subject will receive B regimen in Period 1 and A regimen in Period 2. There will be wash-out period of 5 days between doses.
  Interventions: Drug: RSG XR

INTERVENTIONS:
Drug: RSG XR — RSG XR tablets 8 mg enteric-coated tablet formulation consisting of 3mg fast release plus 5mg slow release. Subject will receive one 8mg of RSG XR on each dosing day. The subject will receive a single oral dose of regiment A or B with 240 milliliter (mL) of water.
  Other Names: BRL-049653

SUMMARY:
The present pharmacokinetic study is designed to compare bioavailability and assess bioequivalence of two Rosiglitazone XR formulations produced at two different sites.Both formulations will be tested in fasting healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18-55 years.
* BMI between 19 - 30 kg/m2

Exclusion criteria:

* Liver function tests above the upper limit
* Excessive alcohol consumption history
* History of Cigarette smoking
* Positive HIV, Hep B or C test
* Positive pregnancy test
* History of heparin sensitivity
* History of glucose intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03-21 (Actual); Primary Completion 2007-05-02 (Actual); Study Completion 2007-05-02 (Actual)

PRIMARY OUTCOMES:
PK samples | at Pre-dose,0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events, vital signs clinical laboratory measurements. | Up to 32

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Neuss, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Results for study AXR107453 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/AXR107453?search=study&search_terms=AXR107453#rs